CLINICAL TRIAL: NCT04799873
Title: Individual Treatment of COVID-19 by Application of Alpha-1-antitrypsin
Brief Title: Alpha-1-Antitrypsin-Deficiency in COVID-19
Acronym: CORSAAR-AAT
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Robert Bals, Professor, Universität des Saarlandes
Other Study IDs: CORSAAR-AAT-001
Record Dates: First submitted 2021-03-14; First posted 2021-03-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — alpha 1-antitrypsin-leukocyte elastase complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, RNA, DNA, EDTA plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: AAT( Alpha 1 Antitrypsin) — AAT administration based on clinical indication
  Other Names: AAT administration based on clinical indication

SUMMARY:
The blood concentrations of alpha-1-antitrypsin are monitored during COVID-19. The clinical course of patients that received AAT infusion for clinical indication is monitored.

DETAILED DESCRIPTION:
The blood concentrations of alpha-1-antitrypsin are monitored during COVID-19. The clinical course of patients that received AAT infusion for clinical indication is monitored. Clinical outcomes, blood inflammatory markers, and virus load are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Infection with SARS-COV2
* Age over 18 years

Exclusion Criteria:

* Unability to consent
* Invasive ventilation

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COVID-19 patients without need for invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical course | 3 months
  Disease course such as death, need for ICU treatment, ventilatory support or deterioration are monitored

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bals, Principal Investigator — UDS
Locations (1):
- Saarland University, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: Undecided